CLINICAL TRIAL: NCT00673322
Title: Phase II/Pilot Trial of Second Generation Designer T Cells in Colorectal Cancer
Brief Title: Trial of Second Generation Designer T Cells in Colorectal Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study will be incorporated into another study.
Sponsor: Roger Williams Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 298-04
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; T cells; Gene Transfer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — 99mTc-anti-carcinoembryonic antigen antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gene Modified T Cells (Experimental): Modified T cells
  Interventions: Biological: Gene Modified T Cells

INTERVENTIONS:
Biological: Gene Modified T Cells — One time infusion Modified T-Cells given through a vein in the arm or a catheter over a 30-60 minute period.
  Other Names: Designer T cells; Anti-CEA

SUMMARY:
The purpose of this study is to collect data on the safety and effectiveness of 2nd generation designer T cells in patients with colorectal cancer. Designer T cells are prepared by collecting white blood cells from the participant, and then modifying these cells in the laboratory so that they recognize the tumor antigen (CEA). These modified cells are then given back into the participant so that they can attack and kill tumor cells.

DETAILED DESCRIPTION:
T cells can penetrate virtually every biologic space and have the power to dispose of normal or malignant cells as seen in viral and autoimmune diseases and in the rare spontaneous remissions of cancer. However, T cells are easily tolerized to self or tumor antigens and "immune surveillance" has manifestly failed in every cancer that is clinically apparent. It is the goal of this study to supply the specificities and affinities to patient T cells without regard for their "endogenous" T cell receptor repertoire, directed by antibody-defined recognition to kill malignant cells based on their expression of antigen. We will achieve this by preparing chimeric IgCD28TCR genes in mammalian expression vectors to yield "designer T cells" from normal patient cells. Prior studies in model systems demonstrated that recombinant IgCD28TCR could direct modified T cells to respond to antigen targets with IL2 secretion, cellular proliferation, and cytotoxicity, the hallmarks of an effective, self-sustaining immune response.

It therefore becomes of paramount interest to extend these studies to a human system of widespread clinical relevance to explore the clinical potential of this new technology. The target antigen for these studies is carcinoembryonic antigen (CEA), which is prominently expressed on tumors of the stomach, colon and rectum, breast, pancreas and other sites. Patients receive a single dose of gene-modified autologous T cells on this dose-escalation trial. Doses are 10^9, 10^10 and 10^11 modified T cells. Patients are monitored for safety and response. Patients are on-study for one month after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Must have cancer of the colon or rectum
* Must have metastatic or unresectable locally advanced disease
* Tumor must express CEA by tumor staining or by elevated serum CEA (>10 ng/ml)
* Must have measurable disease radiologically or by physical exam
* Must have failed potentially curative standard therapy
* Must be 18 years of age or older
* Good performance status (PS 0-1)

Exclusion Criteria:

* Requiring systemic steroids
* Serious medical conditions
* Concurrent malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Determine the safety of using modified T cells by documenting the type and severity of any side effects and establishing the Maximum Tolerated Dose (MTD). | 1 Month

SECONDARY OUTCOMES:
Tumor Response | 1 Month
Pharmacokinetics | 1 Month
Pharmacodynamics | 1 Month

CONTACTS AND LOCATIONS:
Overall Officials: Richard P Junghans, PhD, MD, Principal Investigator — Roger Williams Medical Center
Locations (1):
- Roger Williams Medical Center, Providence, Rhode Island, United States